CLINICAL TRIAL: NCT07188571
Title: Observational Study on Gastric Emptying Rate in Patients With Simple Obesity
Brief Title: Observational Study on GER in Patients With Simple Obesity
Status: Completed | Type: Observational
Sponsor: Jing Ma (Other)
Responsible Party: Sponsor-Investigator, Jing Ma, chief physician, RenJi Hospital
Organization: RenJi Hospital (Other)
Other Study IDs: LY 2025-132-A-RE001
Record Dates: First submitted 2025-09-06; First posted 2025-09-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obesity &Amp;Amp; Overweight; Gastric Emptying Time; Type2 Diabetes Mellitus
Keywords: Observational Study
MeSH Terms: conditions — Obesity; Overweight | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- simple obesity: Inclusion criteria were: diagnosis of obesity (BMI ≥28 kg/m²) and/or waist circumference ≥90 cm in men or ≥85 cm in women, or waist-to-hip ratio ≥0.9 in men and ≥0.85 in women; age 18-65 years; willingness to undergo venous blood sampling and gastric emptying scintigraphy without contraindications; and provision of informed consent. Exclusion criteria included: secondary obesity (e.g., hypothyroidism, Cushing's syndrome, polycystic ovary syndrome); severe cardiovascular, cerebrovascular, autoimmune, or metabolic disease; advanced malignancy; history of drugs affecting glucose-lipid metabolism or gastric emptying; pregnancy or lactation; bleeding tendency; inability to complete venous sampling; contraindications to scintigraphy (such as acute gastrointestinal bleeding, obstruction, perforation, or allergy to test meal) ; refusal of required procedures or consent; and any condition deemed unsuitable.
  Interventions: Diagnostic Test: Gastric emptying scintigraphy

INTERVENTIONS:
Diagnostic Test: Gastric emptying scintigraphy — To assess gastric emptying rates in patients with simple obesity and diagnose the presence of gastric motility abnormalities.
  Other Names: Oral Glucose Tolerance Test (OGTT); Magnetic Resonance Imaging of Fat Distribution

SUMMARY:
Dear Patients, The investigators invite participants to take part in an observational study on gastric emptying rate in individuals with simple obesity. This study has been reviewed and approved by the Ethics Committee of Renji Hospital, affiliated with Shanghai Jiao Tong University School of Medicine. It will be conducted at Renji Hospital and is expected to enroll approximately 100 voluntary participants.

Obesity has become a major global public health challenge. In 2020, an estimated 2.2 billion adults-42% of the global adult population-were affected by overweight and obesity. This number is projected to increase to 3.3 billion by 2035, representing 54% of adults worldwide. Obesity significantly compromises health and is associated with a range of metabolic disorders, including insulin resistance, atherogenic dyslipidemia (characterized by elevated triglycerides and low HDL cholesterol), nonalcoholic fatty liver disease (NAFLD), beta-cell dysfunction, prediabetes, and type 2 diabetes, all of which may lead to serious complications, disability, and premature death.

Gastric emptying refers to the process by which food moves from the stomach into the duodenum. This process is essential for nutrient absorption and is regulated by gastric motility, as well as by neural and hormonal feedback mechanisms mediated by the interaction of nutrients with the small intestine. The rate of gastric emptying determines the pace at which nutrients reach the intestine and influences the enteral nutrient load. It also plays a bidirectional role in regulating blood glucose levels. Therefore, abnormal gastrointestinal motility may represent an important pathophysiological mechanism underlying insulin resistance and impaired glucose tolerance in obese individuals.

To date, most studies on gastric emptying have focused on individuals with diabetes. However, as obesity itself is a major risk factor for metabolic diseases such as type 2 diabetes, further investigation into the distribution patterns of gastric emptying rates in individuals with simple obesity-and its associations with glucose and lipid metabolism, insulin resistance-could provide valuable insights. These insights may support improved diagnosis, risk stratification, and management of obesity-related metabolic disorders, as well as inform the evaluation of weight-loss interventions.

The aim of this study is to assess gastric emptying velocity in patients with simple obesity and to explore its relationship with glucose and lipid metabolic indicators.

This information sheet is intended to help participants decide whether they are willing to allow the use of their historical medical data for research and analysis. Participation in this study is entirely voluntary, and participants' decision will not affect their access to medical care or any of their rights as patients at Renji Hospital. Please be assured that, should participants choose to participate, the investigators will make every effort to protect their safety, privacy, and legal rights throughout the study, in full compliance with applicable ethical and legal standards.

The investigators kindly ask participants to read this notice carefully. If participants have any questions or concerns, they are encouraged to speak with the investigator responsible for explaining the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria for obesity (BMI ≥ 28 kg/m²) and/or waist circumference ≥ 90 cm in adult males, ≥ 85 cm in adult females, or waist-to-hip ratio ≥ 0.9 in males and ≥ 0.85 in females;
* Age 18-65 years;
* Consent to undergo venous blood sampling and gastric emptying scintigraphy, with no contraindications to these procedures;
* Consent to participate in this research project.

Exclusion Criteria:

* Diagnosed with secondary obesity, such as hypothyroidism, Cushing's syndrome, polycystic ovary syndrome, etc.;
* Severe cardiovascular or cerebrovascular disease, rheumatic or immune-mediated disorders;
* Severe metabolic disorders, such as diabetic ketoacidosis, hyperosmolar hyperglycaemic state, etc.;
* Advanced malignant tumours;
* History of medication known to affect glucose/lipid metabolism or gastric emptying rate, such as GLP-1 receptor agonists, glucocorticoids, antibiotics, anxiolytics or antidepressants;
* Pregnancy or lactation;
* Severe bleeding tendency or inability to undergo venous blood sampling;
* Contraindications for gastric emptying scintigraphy, including pregnancy, lactation, severe gastrointestinal disorders such as acute gastrointestinal haemorrhage, intestinal obstruction or perforation, or allergy to components of the test meal;
* Patients refusing gastric emptying scintigraphy, or refusal to sign the informed consent form;
* Other circumstances deemed unsuitable for the study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants included in the study were diagnosed with obesity, aged 18-65 years, without severe wasting diseases, who had not received medication affecting gastric motility, and who had no contraindications for gastric emptying scintigraphy or blood sampling.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
gastric half-emptying time | Baseline
  Gastric half-emptying time (T½) was used as a quantitative parameter to assess gastric emptying function. T½ was defined as the time required for 50% of the ingested standardized radiolabeled test meal to empty from the stomach. Measurement was performed by gastric emptying scintigraphy, during which serial anterior and posterior images were acquired to monitor the time-activity curve of gastric radioactivity. The half-emptying time was determined as the point at which gastric counts declined to 50% of baseline values. Prolongation of T½ is indicative of delayed gastric emptying, commonly observed in conditions such as diabetic gastroparesis or functional dyspepsia, whereas shortening of T½ suggests accelerated gastric emptying, which may occur in certain postoperative states or functional gastrointestinal disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Ren Ji Hospital, Shanghai, Pudong New Area, China

IPD SHARING:
Plan to Share IPD: Undecided
Collaborators to be determined